CLINICAL TRIAL: NCT00187811
Title: Randomised Controlled Trial of Adjuvant Photodynamic Therapy to Reduce Restenosis After Percutaneous Transluminal Angioplasty to the Superficial Femoral Angioplasty
Brief Title: The Safety and Efficacy of Photodynamic Therapy for Femoral Artery Stenosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: UCL/UCLH Clinical Research and Development Fund (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 00/0139
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-09

CONDITIONS: Atherosclerotic Narrowing of the Superficial Femoral Artery; Atherosclerotic Occlusion of the Superficial Femoral Artery
Keywords: Angioplasty,; Restenosis,; Photodynamic therapy

INTERVENTIONS:
Procedure: Delta amino leavulinic acid photodynamic therapy

SUMMARY:
Rstenosis is common after angioplasty of atherosclerotic disease of the femoral artery. Pilot study data suggests that adjuvant photodynamic therapy, using delta amino kleavulinic acid as a photosensitiserr is feasible and safe. This study will examine safety in a larger population and,if recruitment numbers allow, efficacy will be assessed.

Hypothesis:

ALA photodynamic therapy is safe and well tolerated as an adjuvant to angioplasty as a treatment for femoral artery atherosclerotic stenosis or occlusion. A secondary endpoint will be sought : hypothesis : PDT will reduce in restenosis rates following adjuvant photodynamic therapy compared with standard balloon angioplasty in the treatment of superficial femoral arterial disease.

DETAILED DESCRIPTION:
Background:

Percutaneous Transluminal Angioplasty (PTA) is well recognised as a treatment for obstructive vascular disease. Despite an initial high procedural success the technique is limited by the subsequent development of restenosis in up to 50% of patients between 3 and 6 months. ,

The pathological hallmark of restenosis has long been considered to be the development of neointimal hyperplasia consisting of smooth muscle cells and extracellular matrix. We now realise however that both elastic recoil of the vessel and the concept of remodelling are important in determining the overall response of the vessel to injury. Remodelling involves a geometric change in the vessel such that the maximum arterial dimension may increase (positive remodelling) or decrease (negative remodelling). , ,

Despite extensive research no pharmacological or interventional strategy has been shown to have an overwhelming effect on restenosis rates after angioplasty. Recently attention has been focused on the potential of intraluminal radiation therapy (Brachytherapy) and whilst this technique has shown considerable promise there are concerns regarding the long term complications and safety of the ionising radiation for non-malignant disease with reports of vessel wall damage after treatment. ,

Photodynamic therapy is a novel technique that involves the activation of a previously administered photosensitising agent by non thermal laser light. This results in the generation of reactive oxidative products with resulting tissue effects. It is a technique that has been used in the treatment of a variety of malignancies but the realisation that it may influence the response of the vessel wall after balloon injury has been particularly promising. 5 Aminolaevulinic acid (ALA) is a relatively new photosensitising agent which is converted to an active metabolite, Protoporphyrin IX (PPIX) in the biosynthesis of haem. In small animal models photodynamic therapy has been shown to cause medial smooth muscle cell depletion and to reduce the degree of neointimal hyperplasia after injury with no detrimental effects on the mechanical integrity of the vessel wall. , Large animal work using a swine model has confirmed these findings and has also demonstrated that favourable vessel wall remodelling occurs after PDT. Repopulation of the media with smooth muscle cells, after early depletion, has also been demonstrated which is likely to be important when we consider the long term effects of this treatment on the vessel wall.

The use of a large animal model enabled the development of an endovascular system for the delivery of laser light. As a result, and in the light of the findings from large animal studies, it has now been possible to conduct a pilot clinical study looking at the safety and efficacy of adjuvant PDT in patients undergoing repeat PTA for superficial femoral artery (SFA) disease who had restenosed less than 6 months after an earlier angioplasty. In this study it was shown that all patients were asymptomatic 6 months after the procedure with adjuvant PDT there were no arterial or procedural complications. These findings were supported by improvements in non-invasive endpoints and the abscence of significant restenosis as assessed by digital subtraction angiography.

These results were encouraging and we are now in a position to conduct a randomised clinical trial looking at standard balloon angioplasty with and without adjuvant photodynamic therapy in the treatment of peripheral vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of claudication suggested by preliminary Duplex study to be due to superficial femoral artery stenosis or occlusion

Exclusion Criteria:

* Previous surgical graft to superficial femoral artery Known liver dysfunction Previous history of photosensitivity

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2001-02; Study Completion 2006-06

PRIMARY OUTCOMES:
Death
Procedural complications (occlusion, haematoma)
Arterial complications: aneursym, thrombus
Surgical revascularisation (Emergency/Elective)
Repeat PTA
Limb loss

SECONDARY OUTCOMES:
Reccurence of claudication
> 50% loss of initial lumen gain on duplex scanning
PSVR > 2.0
Fall in ABPI
Measured Pre procedure, at 24h then at 1, 3 and 6 months.
A final follow up is planned at 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean R McEwan, MB ChB FRCP, Principal Investigator — University College, London; Stephen Bown, PhD FRCP, Study Director — University College, London
Locations (1):
- University College London NHS Foundation Trust, London, United Kingdom